CLINICAL TRIAL: NCT06993207
Title: Validation of a Home-use Instrument for the Quantification of Cognitive Function in a Population at Risk of Dementia
Brief Title: HOme-based Brain Monitoring With a GARment-EEG to Study Cognitive Decline in the Aging Population
Acronym: Hogar
Status: Recruiting | Type: Observational
Sponsor: Bitbrain (Industry)
Collaborators: Hospital Miguel Servet (Other); Hospital Provincial Nuestra Señora de Gracia (Unknown); Hospital Clínico Zaragoza (Unknown); Universidad de Zaragoza (Other); Instituto de Investigación Sanitaria de Aragón (Unknown)
Responsible Party: Sponsor
Other Study IDs: PI23/373
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Dementia; Mild Cognitive Impairment; Dementia Alzheimers; Dementia, Mixed; Subjective Cognitive Decline; Dementia, Vascular
Keywords: Dementia; MCI; Memory; cognitive decline; EEG; Sleep EEG
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Alzheimer Disease; Mixed Dementias; Dementia, Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Mild Dementia: Patients diagnosed with mild-grade dementia. These individuals will have been diagnosed by a primary care or specialized care physician, following objective clinical criteria: GDS 4 or CDR 1. Dementias in moderate and severe grades (GDS 5-7) will be excluded. Within this group, individuals diagnosed with Alzheimer's dementia, vascular dementia, or mixed dementia will be included. Any other type of dementia will be excluded.
  Interventions: Device: Home Lab
- Mild Cognitive Impairment: Patients diagnosed with mild cognitive impairment. These individuals will have been diagnosed by a primary care or specialized care physician, following objective clinical criteria: GDS 3 or CDR 0.5.
  Interventions: Device: Home Lab
- Subjective Cognitive Decline: Individuals who report subjective memory complaints and do not show objective impairment on cognitive tests. These individuals will have visited their primary care physician claiming memory complaints lasting more than 6 months, but after a standard evaluation, they do not exhibit values within the range compatible with a mild cognitive impairment diagnosis. These individuals correspond to GDS 2 or CDR 0.
  Interventions: Device: Home Lab
- No impairment: Individuals without cognitive alteration. This control group, composed of individuals who are relatives of people belonging to any of the other groups or recruited through advertisements, corresponds to GDS 1 or CDR 0.
  Interventions: Device: Home Lab

INTERVENTIONS:
Device: Home Lab — The main goal is to comprehensively assess the cognitive and behavioral status of all participants, regardless of their assigned groups. Validated clinical tests (considered the gold standard) will be used, with measurements taken at participants' homes using a biosignal monitoring kit-the focal tool of the project. Whether in the control or specific groups, all participants will undergo an identical battery of tests in both the laboratory and home settings. The study design includes an introductory session for participants to understand the study's purpose and sign informed consent. Following consent, participants will have three sessions within a 3 to 6-week timeframe: one for autonomous technology use instruction and the other two for cognitive and functional evaluations.

SUMMARY:
This study will investigate the validity of the HOGAR EEG/PSG monitoring kit designed by Bitbrain as a tool for characterizing and assessing cognitive function in older adults, as well as for detecting and predicting cognitive decline. The kit consists of two EEG headbands and a mobile computing device that allows measurements of sleep patterns (PSG) and brain activity (EEG) in a home environment.

DETAILED DESCRIPTION:
The sample includes 500 participants with various degrees of cognitive impairment according to standard clinical criteria, confirmed through an assessment of cognitive status in the laboratories of Bitbrain and the Miguel Servet Hospital in Zaragoza. This assessment includes an introductory session to the study and two cognitive assessment sessions lasting approximately 2 hours each. The first session includes the explanation of the study protocol, the signing of the informed consent, a short cognitive evaluation using screening tests, and the acquisition of blood samples. The second session includes a recording of brain activity using a versatile semi-dry EEG device (Bitbrain, Spain) under resting conditions and the second part of the battery of cognitive evaluations. During the second session, the battery of cognitive and behavioral tests will be completed.

Outside the hospital environment, participants will receive an in-person tutorial and then take the HOGAR biosignal acquisition kit home for 2 days to collect physiological activity in their daily environment. Each day, they will record EEG in resting conditions and PSG during sleep, both self-administered or with the assistance of a family member. This includes the use of the devices Ikon and Ikon Sleep (Bitbrain, Spain) with a Microsoft Surface with user-friendly software.

This cross-sectional study will allow for the examination of correlations between EEG and PSG acquired in participants' homes with all standard tests in a laboratory setting (especially tests for cognitive decline analysis), and specifically their predictive capacity using artificial intelligence tools. Subsequently, a longitudinal follow-up will explore the possibility of predicting cognitive and behavioral decline based on biosensor measurements in the home environment.

ELIGIBILITY:
General Inclusion Criteria:

* Native Spanish speaker.
* Agree to the examination procedures and tests.
* Ability to involve a close family member or friend for functional evaluation.
* Normal or corrected-to-normal color vision.
* No medical condition requiring chronic systemic medication with psychoactive effects causing confusion.
* No severe psychiatric (according to DSM-V) or neurological diseases (epilepsy with frequent seizures (>1/month) in the last year, multiple sclerosis, etc.).
* No diseases that may interfere with cognitive functions (renal insufficiency on hemodialysis, liver cirrhosis, chronic pulmonary disease with oxygen therapy, solid organ transplant, fibromyalgia, active cancer under treatment).
* No severe hearing and/or visual impairments, neurodevelopmental, or psychomotor disorders.
* No brain injuries that may interfere with cognitive functions (history of traumatic brain injury with parenchymal injury or macroscopic ischemic stroke of large extra-axial vessels or hemorrhagic stroke, brain surgery, brain tumors, or other causes that could result in acquired brain damage such as brain chemotherapy or radiotherapy).
* No treatment with antipsychotic agents in the 6 months prior to the initial assessment.
* No medical condition requiring chronic systemic medication with psychoactive effects causing confusion. No psychiatric or neurological medication.
* No alcohol or drug abuse.
* No serious health problems in the last 12 months (especially neurological or cardiac disorders).

Inclusion Criteria 'Mild Dementia' group:

* Diagnosis of Alzheimer's type dementia, based on a clinical and cognitive assessment conducted by a physician.
* Diagnosis of vascular or mixed type dementia, based on a clinical and cognitive assessment conducted by a physician.
* Lack of autonomy in: 1. basic activities according to the Barthel Index; 2. instrumental activities according to the Lawton Index. Both indices assess dependence associated with the diagnosis of dementia, distinguishing it from the diagnosis of mild cognitive impairment.

Inclusion Criteria 'Mild Cognitive Impairment' group:

* Diagnosis of mild cognitive impairment, based on a clinical and cognitive assessment conducted by a physician.
* Preserved autonomy in: 1. basic activities according to the Barthel Index; 2. instrumental activities according to the Lawton Index. Both indices assess dependence associated with the diagnosis of dementia, distinguishing it from the diagnosis of mild cognitive impairment

Inclusion Criteria 'Subjective Cognitive Decline' group:

* Adherence to SCD-I criteria.
* Attendance at primary care consultation with memory complaints lasting more than 6 months.
* Absence of a diagnosis of mild cognitive impairment or dementia.
* Onset of subjective cognitive decline in the last 5 years.
* Concerns related to subjective cognitive decline (not associated with an acute event) expressed by the participant and/or an informant.
* Cognitive performance within the normal range on cognitive tests (MMSE (Mini Mental State Exam) < 26 / MIS (Memory Impairment Screen) < 6).
* No severe depressive symptoms, indicated by scores > 17* on the 30-item Geriatric Depression Scale.

Inclusion criteria No impairment group:

* Cognitive performance within the normal range on cognitive tests (MMSE < 26 / MIS < 6).
* Absence of a diagnosis of mild cognitive impairment or dementia.
* Not meeting the criteria for SCD-I [21].
* Independent person living in their own home.
* No subjective memory complaints.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our goal is to assemble a diverse sample representing different cognitive impairment levels to validate our developed home kit for effective quantification and prediction of decline. The sample comprises four groups categorized by cognitive level, aiming for gender and age balance.
  1. MILD DEMENTIA: Diagnosed individuals (150) with mild dementia (GDS 4 or CDR 1). Moderate and severe cases (GDS 5-7) are excluded, including Alzheimer's, vascular, or mixed dementia.
  2. MILD COGNITIVE IMPAIRMENT: Diagnosed patients (150) with mild cognitive impairment (GDS 3 or CDR 0.5).
  3. SUBJECTIVE COGNITIVE DECLINE: Individuals reporting memory complaints (100) without objective impairment (GDS 2 or CDR 0).
  4. NO IMPAIRMENT: Individuals without cognitive issues (100), serving as a control group (GDS 1 or CDR 0). Balanced recruitment from family members or advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Validation of HoGar | 1 year
  Validation of an Instrument for Objective and Automated Quantification of Cognitive Function in Older Adults Using Devices for Autonomous Home Use.

SECONDARY OUTCOMES:
Identification of Diagnostic Patterns for Cognitive Impairment Severity Using Home Biosignal Measures. | 1 year
  Utilizing Home Biosignal Measures to Identify Patterns for the Diagnosis of Cognitive Impairment (Including Severity), Distinguishing Them from Those Without Cognitive Impairment (Concurrently Testing the Instrument's Validity).
Predictive Identification of Cognitive Decline and Transitions Using Home Biosignal Measures and Longitudinal Health Data | 1 year
  Identification of Patterns Using Home Biosignal Measures and Longitudinal Health Data to Predict Cognitive Decline and Transitions from Mild Cognitive Impairment to Moderate/Severe Cognitive Impairment or Dementia (Testing the Predictive Validity of the Instrument)

CONTACTS AND LOCATIONS:
Locations (1):
- Bitbrain, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prichep LS, John ER, Ferris SH, Reisberg B, Almas M, Alper K, Cancro R. Quantitative EEG correlates of cognitive deterioration in the elderly. Neurobiol Aging. 1994 Jan-Feb;15(1):85-90. doi: 10.1016/0197-4580(94)90147-3. PMID 8159266
- [Background] Prichep LS, John ER, Ferris SH, Rausch L, Fang Z, Cancro R, Torossian C, Reisberg B. Prediction of longitudinal cognitive decline in normal elderly with subjective complaints using electrophysiological imaging. Neurobiol Aging. 2006 Mar;27(3):471-81. doi: 10.1016/j.neurobiolaging.2005.07.021. Epub 2005 Oct 6. PMID 16213630